CLINICAL TRIAL: NCT07240675
Title: A Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Doses of KLA478 in Healthy Volunteers
Brief Title: Single-dose,First-in-human of KLA478
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hunan Kelun Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KLA478-101
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers
Keywords: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- pramipexole hydrochloride sustained-release tablets 0.375mg (Active Comparator): 10 volunteers receive pramipexole hydrochloride sustained-release tablets 0.375mg
  Interventions: Drug: pramipexole hydrochloride sustained-release tablets
- KLA478 2mg (Experimental): 8 volunteers receive KLA478 2mg，2 volunteers receive the same volume placebo
  Interventions: Drug: KLA478; Drug: placebo
- KLA478 5mg (Experimental): 8 volunteers receive KLA478 5mg，2 volunteers receive the same volume placebo
  Interventions: Drug: KLA478; Drug: placebo
- KLA478 10mg (Experimental): 8 volunteers receive KLA478 10mg，2 volunteers receive the same volume placebo
  Interventions: Drug: KLA478; Drug: placebo

INTERVENTIONS:
Drug: pramipexole hydrochloride sustained-release tablets — P.O., single dose
  Arms: pramipexole hydrochloride sustained-release tablets 0.375mg
Drug: KLA478 — intramuscular injection, single dose
  Arms: KLA478 10mg; KLA478 2mg; KLA478 5mg
Drug: placebo — intramuscular injection, single dose
  Arms: KLA478 10mg; KLA478 2mg; KLA478 5mg

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability and pharmacokinetics of single doses of KLA478 in healthy volunteers；

DETAILED DESCRIPTION:
This study is a single-center, randomized/non-randomized, single ascending dose（SAD）, Phase I clinical trial conducted in healthy subjects, divided into two parts:

Part 1 is an open-label single-dose study of active comparator to evaluate the pharmacokinetic characteristics of active comparator in healthy subjects； Part 2 is a randomized, double-blind, placebo-controlled single ascending dose study of KLA478: The purpose of this study is to evaluate the safety and tolerability and pharmacokinetics of single doses of KLA478 in healthy volunteers；

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form
2. Health participants (Age: 18~45 years);
3. Body Weight: Male≥50.0kg, Female≥45.0kg; 19 ≤BMI≤ 28.0kg/m2;
4. Clinical examination normal, or abnormal with no clinical significance；
5. Agreed to use contraception for 3-6 months.

Exclusion Criteria:

1. Allergy or Drug hypersensitivity;
2. Clinically significant Medical History；
3. Subjects with difficult venous blood collection/intolerance to venipuncture, or with a history of needle phobia/blood phobia；
4. Assess injection site abnormalities；
5. History of drugs that may interact with pramipexole within 1 month；
6. History of any Medication within 2 weeks；
7. Massive blood loss (> 200 mL) in the past 3 months；
8. History of any surgery within 3 months, or plan to undergo surgery during the trial；
9. History of any clinical study within 90 days；
10. History of any vaccine within 1 month，or Plan to get vaccinated during the trial period；
11. systolic blood pressure decreased ≥20 mmHg or diastolic blood pressure decreased ≥10 mmHg within 3 minutes from supine to upright position；
12. QTcF>450 ms；
13. Abnormal vital signs with clinical significance ；
14. Serum potassium level exceeds the reference range.；
15. Pre-transfusion test abnormal；
16. Lactation or pregnancy test positive ；
17. History of any drug abuse or positive drugs of abuse test result；
18. Previous alcohol abuse or unwillingness to stop drinking or alcohol breath test positive；
19. more than 3 cigarettes per day in 3 months, or unwilling to stop during the trial；
20. Intake of special diets that affect drug absorption, distribution, metabolism and excretion within 48 hours；
21. Have special requirements for diet；
22. Unprotected sexual behavior within 2 weeks;
23. engaged in driving vehicles, operating machinery, high-altitude work or other potentially dangerous behavior;
24. Inappropriate for participation in this trial as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-26 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Up to Day 109

SECONDARY OUTCOMES:
PK parameter Tmax | up to Day 90
  Time of Cmax (Tmax) after single dose
PK parameter Cmax | up to Day 90
  Maximum peak plasma concentration (Cmax) after single dose
PK parameter AUC0-t | up to Day 90
  Area under the concentration-time curve (AUC0-t) from time zero to time "t" after single dose
PK parameter AUC0-∞ | up to Day 90
  AUC from time zero to infinity (AUC0-∞) after single dose
PK parameter AUC_%Extrap | up to Day 90
  Area Under the Curve Percent Extrapolated
PK parameter Tlast | Area Under the Curve Percent Extrapolated
  Time of Last measurable concentration
PK parameter λz | up to Day 90
  Elimination Rate Constant
PK parameter t1/2 | up to Day 90
  Terminal-phase elimination half-life (t1/2) after single dose
PK parameter CL/F | up to Day 90
  Clearance adjusted for bioavailability
PK parameter Vz/F | up to Day 90
  Volume of Distribution adjusted for bioavailability
PK parameter MRT | up to Day 90
  Mean Resident Time

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No